CLINICAL TRIAL: NCT06226168
Title: Effect of the Author's Training Program in Normobaric Hypoxia on Changes in Bone Turnover Markers and Carbohydrate and Lipid Metabolism in Premenopausal Women
Brief Title: Effects of Normobaric Hypoxia Exercise Program on Bone Turnover Markers and Metabolism in Premenopausal Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University School of Physical Education, Krakow, Poland (Other)
Collaborators: Ministry of Education and Science,Poland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NdS-II/SP/0512/2023/01
Record Dates: First submitted 2023-12-11; First posted 2024-01-26 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Hypoxia
Keywords: bone turnover; carbohydrate metabolism; lipid metabolism; normobaric hypoxia
MeSH Terms: conditions — Hypoxia | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (No Intervention): The control group will not undergo the training program.
- Training in normobaric hypoxia (Experimental): Training performed under normobaric hypoxia (Week I-1600m above sea level; Week II-1800m above sea level; Week III-2200m above sea level; Week IV-2600m above sea level) and thermoneutral conditions (21°C) and constant humidity (40%).
  Interventions: Other: exercise and environmental conditions
- Training in normoxia (Experimental): Description: Training performed in normoxia (223 m above sea level) and thermoneutral conditions (21°C) and constant humidity (40%).
  Interventions: Other: exercise and environmental conditions
- Passive exposure to normobaric hypoxia (Experimental): Passive exposure to normobaric hypoxia conditions (Week I -1600m above sea level; Week II -1800m above sea level; Week III -2200m above sea level; Week IV-2600m above sea level) and thermoneutral conditions (21°C) and constant humidity (40%).
  Interventions: Other: exercise and environmental conditions

INTERVENTIONS:
Other: exercise and environmental conditions — Participants will perform endurance-strength training for 4 weeks in a variety of environmental conditions. Somatic indices and quantitative indicators of bone mass (bone mineral density) will be measured both before and after the training period. Before the first training day and the day after the last training day, blood will be drawn for biochemical analysis.
  Arms: Training in normobaric hypoxia; Training in normoxia
Other: exercise and environmental conditions — Passive exposure to normobaric hypoxia conditions. No training intervention. There will be a measurement of selected somatic indices and a quantitative measurement of bone mass indices (bone mineral density). A blood draw for biochemical analysis will be performed.
  Arms: Passive exposure to normobaric hypoxia

SUMMARY:
The impact of a proprietary training program in normobaric hypoxia on changes in bone turnover markers as well as carbohydrate and lipid metabolism in premenopausal women falls within the realm of physical culture for an active and healthy society. Within this context, the implementation of a project is supported aiming to:

1. Monitor, support, and promote physical development, fitness, and physical activity in society, by assessing the effects of a proprietary training program in normobaric hypoxia on changes in bone turnover markers as well as carbohydrate and lipid metabolism in premenopausal women.
2. Develop and implement innovative methods, forms, and means of physical activation and training for individuals of various ages, by formulating general assumptions of an endurance-strength training concept under normobaric hypoxia conditions, concerning changes in bone turnover markers as well as carbohydrate and lipid metabolism in premenopausal women.
3. Prevent injuries in physical education and sports, by designing a useful training program for osteoporosis prevention as well as for managing carbohydrate and lipid metabolism disorders in premenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* No significant cardiovascular, respiratory system diseases and musculoskeletal system,
* No contraindications to physical activity. ECG, baseline urinalysis, morphology are required.
* T-score within normal limits (+1.0 to -1.0).
* Informed consent of the patient to participate in the study.

Exclusion Criteria:

* Use of hormone replacement therapy (HRT).
* Use of substances (cigarettes, alcohol).
* Any training (including hypoxia training or exposure) performed in the 6 months prior to the beginning of the intervention
* Any other factors determined by the study investigators as unsuitable for participation.

Ages: 50 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Blood analysis- part 1 | Before (10 minutes) and after (3 minutes) the first and last training.The training will last 4 weeks and will consist of 12 workouts
  Bone turnover markers: bone-specific alkaline phosphatase (ng/ml), osteocalcin (ng/ml), N-terminal telopeptide of type I collagen (ng/ml), osteoprotegerin (ng/ml), 25-hydroxyvitamin D3 metabolite (ng/ml).
Blood analysis- part 2 | Before (10 minutes) and after (3 minutes) the first and last training.The training will last 4 weeks and will consist of 12 workouts
  Hormones of lipid metabolism: adiponectin (μg/mL)
Blood analysis- part 3 | Before (10 minutes) and after (3 minutes) the first and last training.The training will last 4 weeks and will consist of 12 workouts
  Hormones of lipid metabolism: lipid profile (mg/dL)
Blood analysis- part 4 | Before (10 minutes) and after (3 minutes) the first and last training.The training will last 4 weeks and will consist of 12 workouts
  Hormones of lipid metabolism: lipoprotein atherogenicity index (no unit)
Blood analysis- part 5 | Before (10 minutes) and after (3 minutes) the first and last training.The training will last 4 weeks and will consist of 12 workouts
  Hormones of carbohydrate metabolism: glucose (mg/dL)
Blood analysis- part 6 | Before (10 minutes) and after (3 minutes) the first and last training.The training will last 4 weeks and will consist of 12 workouts
  Hormones of carbohydrate metabolism: insulin (IU/mL), leptin (IU/mL), ghrelin (IU/mL)
Blood analysis- part 7 | Before (10 minutes) and after (3 minutes) the first and last training.The training will last 4 weeks and will consist of 12 workouts
  Thyroid hormones: Thyroid Stimulating Hormone (IU/L)
Blood analysis- part 8 | Before (10 minutes) and after (3 minutes) the first and last training.The training will last 4 weeks and will consist of 12 workouts
  Vitamins: Vitamin D (ng/mL)
Blood analysis- part 9 | Before (10 minutes) and after (3 minutes) the first and last training.The training will last 4 weeks and will consist of 12 workouts
  Plasma volume changes (ml/kg)
Blood analysis- part 10 | Before (10 minutes) and after (3 minutes) the first and last training.The training will last 4 weeks and will consist of 12 workouts
  Rheology: viscosity (Pa·s), viscoelasticity (Pa·s)
Blood analysis- part 11 | Before (10 minutes) and after (3 minutes) the first and last training.The training will last 4 weeks and will consist of 12 workouts
  Rheology: shear rate (s-¹)
Blood analysis- part 12 | Before (10 minutes) and after (3 minutes) the first and last training.The training will last 4 weeks and will consist of 12 workouts
  Rheology: shear stress (Pa), elastic modulus (Pa)
Blood analysis- part 13 | Before (10 minutes) and after (3 minutes) the first and last training.The training will last 4 weeks and will consist of 12 workouts
  Blood biochemistry: erythrocytes (million/μL)
Blood analysis- part 14 | Before (10 minutes) and after (3 minutes) the first and last training.The training will last 4 weeks and will consist of 12 workouts
  Blood biochemistry: leukocytes (thousand/μL), platelets (thousand/μL)
Blood analysis- part 15 | Before (10 minutes) and after (3 minutes) the first and last training.The training will last 4 weeks and will consist of 12 workouts
  Blood biochemistry: hemoglobin (g/dL)
Blood analysis- part 16 | Before (10 minutes) and after (3 minutes) the first and last training.The training will last 4 weeks and will consist of 12 workouts
  Blood biochemistry: hematocrit (%), red cell distribution width (%)
Blood analysis- part 17 | Before (10 minutes) and after (3 minutes) the first and last training.The training will last 4 weeks and will consist of 12 workouts
  Blood biochemistry: mean corpuscular volume (femtoliter)
Blood analysis- part 18 | Before (10 minutes) and after (3 minutes) the first and last training.The training will last 4 weeks and will consist of 12 workouts
  Blood biochemistry: mean corpuscular hemoglobin (picogram)
Blood analysis- part 19 | Before (10 minutes) and after (3 minutes) the first and last training.The training will last 4 weeks and will consist of 12 workouts
  Blood biochemistry: mean corpuscular hemoglobin concentration (g/dL), albumin (g/dL)
Blood analysis- part 20 | Before (10 minutes) and after (3 minutes) the first and last training.The training will last 4 weeks and will consist of 12 workouts
  Blood biochemistry: creatinine (mg/dL), bilirubin (mg/dL), blood urea nitrogen (mg/dL)
Blood analysis- part 21 | Before (10 minutes) and after (3 minutes) the first and last training.The training will last 4 weeks and will consist of 12 workouts
  Blood biochemistry: erythrocyte sedimentation rate (mm/h)
Blood analysis- part 22 | Before (10 minutes) and after (3 minutes) the first and last training.The training will last 4 weeks and will consist of 12 workouts
  Blood biochemistry: alanine aminotransferase (U/L), aspartate aminotransferase (U/L)
Blood analysis- part 23 | Before (10 minutes) and after (3 minutes) the first and last training.The training will last 4 weeks and will consist of 12 workouts
  Blood biochemistry: ferritin (ng/mL)
Bone mass- part 1 | 1 day before and 1 day after the training program. Training will last 4 weeks.
  To identify quantitative indicators of bone mass, a densitometric study will be performed using dual energy X-ray absorptiometry (DXA). Selected quantitative indicators of bone mass will be measured: bone mineral density (g/cm^2).
Bone mass- part 2 | 1 day before and 1 day after the training program. Training will last 4 weeks.
  To identify quantitative indicators of bone mass, a densitometric study will be performed using dual energy X-ray absorptiometry (DXA). Selected quantitative indicators of bone mass will be measured: T-score (no unit).
Bone mass- part 3 | 1 day before and 1 day after the training program. Training will last 4 weeks.
  To identify quantitative indicators of bone mass, a densitometric study will be performed using dual energy X-ray absorptiometry (DXA). Selected quantitative indicators of bone mass will be measured: Z-score (no unit).
Bone mass- part 4 | 1 day before and 1 day after the training program. Training will last 4 weeks.
  To identify quantitative indicators of bone mass, a densitometric study will be performed using dual energy X-ray absorptiometry (DXA). Selected quantitative indicators of bone mass will be measured: relative skeletal-muscular index (kg/m^2).
Somatic indicators- part 1 | 1 day before and 1 day after the training program. Training will last 4 weeks.
  A densitometry study using dual energy X-ray absorptiometry (DXA) will be conducted to determine body composition: lean body mass (kg).
Somatic indicators- part 2 | 1 day before and 1 day after the training program. Training will last 4 weeks.
  A densitometry study using dual energy X-ray absorptiometry (DXA) will be conducted to determine body composition: percentage of body fat (%).
Somatic indicators- part 3 | 1 day before and 1 day after the training program. Training will last 4 weeks
  A densitometry study using dual energy X-ray absorptiometry (DXA) will be conducted to determine body composition: fat mass (kg).

CONTACTS AND LOCATIONS:
Overall Officials: Małgorzata Bagińska, MSc, Principal Investigator — Student of Doctoral studies, University of Physical Education in Kraków, Poland
Locations (1):
- University School of Physical Education in Cracow, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No